CLINICAL TRIAL: NCT00936013
Title: Antiviral and Chinese Medicinal Herbs Treatment on Novel Influenza A (H1N1) Virus Pneumonia: Multi-centre, Prospective, Randomized Controlled Study
Brief Title: Chinese Medicinal Herbs Treatment on Novel Influenza A (H1N1)Pneumonia: Multi-centre, Prospective, Randomized Controlled Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Wang Chen, Capital Medical University affiliated Beijing Chaoyang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Z09000700090903-2
Record Dates: First submitted 2009-07-08; First posted 2009-07-09 (Estimated); Last update posted 2009-11-02 (Estimated); Status verified 2009-11

CONDITIONS: Influenza
Keywords: novel influenza A(H1N1); chinese medicinal herbs
MeSH Terms: conditions — Influenza, Human | interventions — Oseltamivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- oseltamivir (Experimental): single antiviral treatment
  Interventions: Drug: oseltamivir
- oseltimivir and chinese medicinal herbs (Experimental): combination treatment
  Interventions: Drug: oseltamivir and chinese medicinal herbs

INTERVENTIONS:
Drug: oseltamivir — 75mg p.o Bid for 5 days
  Other Names: Tamiflu
  Arms: oseltamivir
Drug: oseltamivir and chinese medicinal herbs — oseltamivir: 75mg p.o bid for 5 days chinese medicinal herbs:200ml p.o qid for 5 days
  Arms: oseltimivir and chinese medicinal herbs

SUMMARY:
The purpose of the study is to determine whether the combination treatment of Chinese medicinal herbs and oseltamivir is more effective than single oseltamivir in treating novel influenza A (H1N1) pneumonia.

DETAILED DESCRIPTION:
The antiviral agent, oseltamivir, is recommended by the World Health Organization (WHO) to treat recent outbreak novel influenza A (H1N1) virus infection around world. But limited stock and resistant strain emergence raised increasing concerns. Chinese medicinal herbs, are derived from plants and usually incorporate one or more herbs as the basic drug(s) to treat the disease. The investigators performed RCT to indicate that a combination treatment of Chinese medicinal herbs and oseltamivir is more effective than single oseltamivir in treating novel influenza A (H1N1) pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed novel influenza A(H1N1) case with laboratory evidence
* 70 ys ≥ age ≥14ys
* Within 72hr after the onset of symptoms(body temperature≥37.5℃ with at least one respiratory symptom (cough, sore throat, or nasal symptom)
* New lung infiltration showed by chest radiology(x-ray or CT)

Exclusion Criteria:

* Age<14ys or >70ys
* Pregnancy
* Severe chronic underlying diseases: severe COPD(FEV1/EVC <70% and FEV1 <30% predicted or respiratory failure or congestive heart failure), severe liver disfunction（ALT or AST ≥3 times normal elevation), renal disfunction（Cr>2mg/dL), chronic heart failure(NYHA Ⅲ-Ⅳ grade）
* Immunocompromised patients(cancer, organ transplant, AIDS and a history of treatment with immunosuppressive drug and glucocorticoids in the past 3 months)
* Taken Chinese medicinal herbs, antiviral or antibiotic drug in the past 2 weeks
* Inoculation influenza vaccination
* One of the following items appeared at the enrollment

  * respiratory failure：PaO2<60mmHg and/or PCO2>50mmHg or PaO2/FiO2≤300
  * circulation failure: despite adequate fluid resuscitation and cardiac output, systolic <90mmHg or requirement inotropic support
  * renal function failure: despite adequate fluid resuscitation and cardiac output, urine ≤ 0.5ml/kg.h, Cr or BUN≥1 time normal elevation
  * liver function failure: total bilirubin>34μmol/L or ALT/AST ≥3 times normal elevation
* Other unappropriated enrollment situations considered by investigator

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2009-08; Primary Completion 2011-07 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Efficacy rate in 5 days (defined as failure: SaO2<90% at room air or temperature elevated continuously) | two years

SECONDARY OUTCOMES:
Time to resolution of fever(defined as the period from start of study-drug to relief of fever) | two years
Time to resolution of respiratory symptoms(defined as the period from start of study-drug to relief of symptoms) | two years
Virus shedding time | two years
Infiltration resolution of chest radiology | two years
SaO2 and PaO2/FiO2(arterial blood gas) | two years

CONTACTS AND LOCATIONS:
Overall Officials: Chen Wang, Doctor, Study Chair — Beijing Chao Yang Hospital; Qingquan Liu, Docter, Study Director — Beijing Chinese Traditional Medicine University affiliated Dongzhimen Hospital; Yu Mao, Doctor, Study Director — Beijing Ditan Hospital
Locations (1):
- Capital Medical University affiliated Bejing Chaoyang Hospital, Beijing Respiratory Medicine Institute, Beijing, China